CLINICAL TRIAL: NCT02286570
Title: Face-to-face Tracheal Intubation With Fastrach or Videolaryngoscopes
Brief Title: Face-to-face Tracheal Intubation: a Comparison of Airtraq, Glidescope and Fastrach
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: KOU KAEK 2014/255
Record Dates: First submitted 2014-10-31; First posted 2014-11-10 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Intubation Difficult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- face-to-face intubation of Glidescope (Active Comparator): patients were intubated using glidescope by face-to-face approach
  Interventions: Device: Glidescope
- face-to-face intubation with Airtraq (Active Comparator): patients were intubated using the Airtraq by face-to-face approach
  Interventions: Device: Airtraq
- face-to-face intubation with fastrach (Active Comparator): patients were intubated using the Fastrach by face-to-face approach
  Interventions: Device: Fastrach

INTERVENTIONS:
Device: Glidescope — videolaryngoscope used for endotracheal intubation
  Arms: face-to-face intubation of Glidescope
Device: Airtraq — videolaryngoscope used for endotracheal intubation
  Arms: face-to-face intubation with Airtraq
Device: Fastrach — intubating laryngeal mask airway used for blind endotracheal intubation
  Arms: face-to-face intubation with fastrach

SUMMARY:
Trauma victims had to be intubated at the scene of area in different conditions. Face-to-face intubation in an entrapped patient is one of these situations. The investigators want to compare the efficacy of Glidescope, Airtraq and Fastrach in simulating face-ro-face intubation in adult patients aged between 18-60 years.

DETAILED DESCRIPTION:
The investigators record the demographic and the airway data of the patients (thyromental distance, sternomental distance, mallampati score, mandibula protrusions, interincisor distance..etc). The hemodynamic data of the patients baseline preoperatively, after induction, after insertion of the device, after intubation, and 2 minutes intervals after intubation during the ten minutes. Cormack-Lehane grade of the videolaryngoscopes, insertion time, intubation time, need of optimisation maneuvers, mucosal damage, teeth and tongue damage, postoperative sore throat, hoarseness, dysphagia were recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* Elective surgery requiring endotracheal intubation
* Normal airway variables
* BMI< 30

Exclusion Criteria:

* < 18 years or > 60 years
* Emergency procedures
* Known difficult airways
* BMI> 30

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
intubation time | elapsing between the handling of the device till intubation 2 minutes
  2 minutes

SECONDARY OUTCOMES:
mucosal damage | blood on the device after removal 1 minute
  1 minute after removal
postoperative minor complications sore troat, teeth damage, tongue damage, desaturation, hoarseness, disphagia | sore troat, teeth damage, tongue damage, desaturation, hoarseness, disphagia 30 minutes
  30 minutes after extubation
need of optimisation maneuvers | chandy, side-to-side, handling force, up-down, reinserting 15 minutes
  during 15 minutes while intubation
hemodynamic changes (mean arteriial pressure) | entübation and after 15 minutes
  mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Zehra I ARSLAN, Doctor, Principal Investigator — Anesthesiology and Reanimation